CLINICAL TRIAL: NCT00013130
Title: Ambulatory Care Quality Improvement (ACQUIP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: SDR 96-002
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-02

CONDITIONS: Health Status Measures; Outcomes; Continuous Quality Improvement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: Provision of health status information to patients provider

INTERVENTIONS:
Behavioral: Provision of health status information to patients provider

SUMMARY:
Health care organizations, including the VA, are investing substantial effort to improve quality of care. As part of this process, greater emphasis is being placed on measurement of outcomes, and in particular, functional outcomes and satisfaction as reported by patients.

DETAILED DESCRIPTION:
Background:

Health care organizations, including the VA, are investing substantial effort to improve quality of care. As part of this process, greater emphasis is being placed on measurement of outcomes, and in particular, functional outcomes and satisfaction as reported by patients.

Objectives:

ACQUIP was designed to determine whether quality and outcomes of health care improve when primary care providers have access to regular assessments of their patients' health and function along with routine clinical data and information about clinical guidelines.

Methods:

This study was a randomized trial conducted at the General Internal Medicine Clinics of seven VA facilities. Each participating GIMC is organized into discrete firms staffed by different groups of providers who care for different patients. One randomly selected firm received the intervention and one served as control. Patients who made at least one GIMC visit in the last year were eligible to participate. Patients were surveyed at baseline to determine active medical problems. Subsequent mailings included a general evaluation of health status (SF-36), a satisfaction questionnaire and, as appropriate, one of six condition-specific questionnaires: the Seattle Angina Questionnaire, the Seattle Obstructive Lung Disease Questionnaire, the Hopkins Symptom Checklist (depression), and questionnaires regarding diabetes, drinking, and hypertension. Clinical/utilization data were downloaded weekly from VISTA and supplemented with data from Austin. The intervention consisted of multi-faceted reports to patients' primary care providers (at the time of patient visits) showing trended physiologic and health status data and guideline-derived recommendations. Clinicians also received periodical reports displaying trends in the health status and satisfaction of their patients compared with their clinic as a whole. Reports were supplemented by training on QI and health status measures.

Status:

Data collection was completed on April 1, 2000. Analysis of trial results will be completed January, 2001.

ELIGIBILITY:
Inclusion Criteria:

Enrolled in VA GIM clinic with visit in past year

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62487 (Estimated)
Dates: Study Completion 2001-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephan D. Fihn, MD MPH, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA; Kenneth E. Rosenfeld, MD, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA; Marisue Cody, PhD RN MPA, Principal Investigator — Central Arkansas Veterans Healthcare System Eugene J. Towbin Healthcare Center, Little Rock, AR
Locations (5):
- United States (5):
  - Central Arkansas Veterans Healthcare System Eugene J. Towbin Healthcare Center, Little Rock, AR, No. Little Rock, Arkansas
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California
  - White River Junction VA Medical Center, White River Junction, VT, White River Junction, Illinois
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington

REFERENCES:
- [Result] Williams EC, Peytremann-Bridevaux I, Fan VS, Bryson CL, Blough DK, Kivlahan DR, Bradley KA. The association between alcohol screening scores and health status in male veterans. J Addict Med. 2010 Mar;4(1):27-37. doi: 10.1097/ADM.0b013e3181a196b5. PMID 21769021
- [Result] Fan VS, Bridevaux PO, McDonell MB, Fihn SD, Besser LM, Au DH. Regional variation in health status among chronic obstructive pulmonary disease patients. Respiration. 2011;81(1):9-17. doi: 10.1159/000320115. Epub 2010 Aug 17. PMID 20720400
- [Result] Bryson CL, Au DH, Sun H, Williams EC, Kivlahan DR, Bradley KA. Alcohol screening scores and medication nonadherence. Ann Intern Med. 2008 Dec 2;149(11):795-804. doi: 10.7326/0003-4819-149-11-200812020-00004. PMID 19047026
- [Result] Krumholz HM, Anderson JL, Bachelder BL, Fesmire FM, Fihn SD, Foody JM, Ho PM, Kosiborod MN, Masoudi FA, Nallamothu BK; American College of Cardiology/American Heart Association Task Force on Performance Measures; American Academy of Family Physicians; American College of Emergency Physicians; American Association of Cardiovascular and Pulmonary Rehabilitation; Society for Cardiovascular Angiography and Interventions; Society of Hospital Medicine. ACC/AHA 2008 performance measures for adults with ST-elevation and non-ST-elevation myocardial infarction: a report of the American College of Cardiology/American Heart Association Task Force on Performance Measures (Writing Committee to Develop Performance Measures for ST-Elevation and Non-ST-Elevation Myocardial Infarction) Developed in Collaboration With the American Academy of Family Physicians and American College of Emergency Physicians Endorsed by the American Association of Cardiovascular and Pulmonary Rehabilitation, Society for Cardiovascular Angiography and Interventions, and Society of Hospital Medicine. J Am Coll Cardiol. 2008 Dec 9;52(24):2046-99. doi: 10.1016/j.jacc.2008.10.012. No abstract available. PMID 19056000
- [Result] Krumholz HM, Anderson JL, Bachelder BL, Fesmire FM, Fihn SD, Foody JM, Ho PM, Kosiborod MN, Masoudi FA, Nallamothu BK; American College of Cardiology/American Heart Association Task Force on Performance Measures; American Academy of Family Physicians; American College of Emergency Physicians; American Association of Cardiovascular and Pulmonary Rehabilitation; Society for Cardiovascular Angiography and Interventions; Society of Hospital Medicine. ACC/AHA 2008 performance measures for adults with ST-elevation and non-ST-elevation myocardial infarction: a report of the American College of Cardiology/American Heart Association Task Force on Performance Measures (Writing Committee to develop performance measures for ST-elevation and non-ST-elevation myocardial infarction): developed in collaboration with the American Academy of Family Physicians and the American College of Emergency Physicians: endorsed by the American Association of Cardiovascular and Pulmonary Rehabilitation, Society for Cardiovascular Angiography and Interventions, and Society of Hospital Medicine. Circulation. 2008 Dec 9;118(24):2596-648. doi: 10.1161/CIRCULATIONAHA.108.191099. Epub 2008 Nov 10. No abstract available. PMID 19001027
- [Result] Bryson CL, Au DH, Young B, McDonell MB, Fihn SD. A refill adherence algorithm for multiple short intervals to estimate refill compliance (ReComp). Med Care. 2007 Jun;45(6):497-504. doi: 10.1097/MLR.0b013e3180329368. PMID 17515776
- [Result] Parimon T, Chien JW, Bryson CL, McDonell MB, Udris EM, Au DH. Inhaled corticosteroids and risk of lung cancer among patients with chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2007 Apr 1;175(7):712-9. doi: 10.1164/rccm.200608-1125OC. Epub 2006 Dec 21. PMID 17185647
- [Result] DeSalvo KB, Fan VS, McDonell MB, Fihn SD. Predicting mortality and healthcare utilization with a single question. Health Serv Res. 2005 Aug;40(4):1234-46. doi: 10.1111/j.1475-6773.2005.00404.x. PMID 16033502
- [Result] Liu CF, Campbell DG, Chaney EF, Li YF, McDonell M, Fihn SD. Depression diagnosis and antidepressant treatment among depressed VA primary care patients. Adm Policy Ment Health. 2006 May;33(3):331-41. doi: 10.1007/s10488-006-0043-5. PMID 16755394
- [Result] Davis GE, Bryson CL, Yueh B, McDonell MB, Micek MA, Fihn SD. Treatment delay associated with alternative medicine use among veterans with head and neck cancer. Head Neck. 2006 Oct;28(10):926-31. doi: 10.1002/hed.20420. PMID 16755583
- [Result] Spertus JA, McDonell M, Woodman CL, Fihn SD. Association between depression and worse disease-specific functional status in outpatients with coronary artery disease. Am Heart J. 2000 Jul;140(1):105-10. doi: 10.1067/mhj.2000.106600. PMID 10874270
- [Result] Diehr P, Patrick DL, Spertus J, Kiefe CI, McDonell M, Fihn SD. Transforming self-rated health and the SF-36 scales to include death and improve interpretability. Med Care. 2001 Jul;39(7):670-80. doi: 10.1097/00005650-200107000-00004. PMID 11458132
- [Result] Bridevaux IP, Bradley KA, Bryson CL, McDonell MB, Fihn SD. Alcohol screening results in elderly male veterans: association with health status and mortality. J Am Geriatr Soc. 2004 Sep;52(9):1510-7. doi: 10.1111/j.1532-5415.2004.52414.x. PMID 15341553
- [Result] Burman ML, Kivlahan D, Buchbinder M, Broglio K, Zhou XH, Merrill JO, McDonell MB, Fihn SD, Bradley KA; Ambulatory Care Quality Improvement Project Investigators. Alcohol-related advice for Veterans Affairs primary care patients: Who gets it? Who gives it? J Stud Alcohol. 2004 Sep;65(5):621-30. doi: 10.15288/jsa.2004.65.621. PMID 15536772
- [Result] Bradley KA, Kivlahan DR, Zhou XH, Sporleder JL, Epler AJ, McCormick KA, Merrill JO, McDonell MB, Fihn SD. Using alcohol screening results and treatment history to assess the severity of at-risk drinking in Veterans Affairs primary care patients. Alcohol Clin Exp Res. 2004 Mar;28(3):448-55. doi: 10.1097/01.alc.0000117836.38108.38. PMID 15084903
- [Result] Fan VS, Burman M, McDonell MB, Fihn SD. Continuity of care and other determinants of patient satisfaction with primary care. J Gen Intern Med. 2005 Mar;20(3):226-33. doi: 10.1111/j.1525-1497.2005.40135.x. PMID 15836525
- [Result] Tu SP, McDonell MB, Spertus JA, Steele BG, Fihn SD. A new self-administered questionnaire to monitor health-related quality of life in patients with COPD. Ambulatory Care Quality Improvement Project (ACQUIP) Investigators. Chest. 1997 Sep;112(3):614-22. doi: 10.1378/chest.112.3.614. PMID 9315792
- [Result] Kiefe CI, McDonell MB, Martin D, Fihn S. Patient satisfaction and perceived health status: general and coronary artery disease specific racial differences among veterans [abstract]. [Abstract]. Abstract book / Annual Meeting. Association for Health Services Research. Meeting. 1997 Oct 15; 14P70:70.
- [Result] Au DH, Udris EM, Curtis JR, McDonell MB, Fihn SD; ACQUIP Investigators. Association between chronic heart failure and inhaled beta-2-adrenoceptor agonists. Am Heart J. 2004 Nov;148(5):915-20. doi: 10.1016/j.ahj.2004.03.048. PMID 15523327
- [Result] Au DH, Bryson CL, Fan VS, Udris EM, Curtis JR, McDonell MB, Fihn SD. Beta-blockers as single-agent therapy for hypertension and the risk of mortality among patients with chronic obstructive pulmonary disease. Am J Med. 2004 Dec 15;117(12):925-31. doi: 10.1016/j.amjmed.2004.07.043. PMID 15629731
- [Result] Spertus JA, Winder JA, Dewhurst TA, Deyo RA, Fihn SD. Monitoring the quality of life in patients with coronary artery disease. Am J Cardiol. 1994 Dec 15;74(12):1240-4. doi: 10.1016/0002-9149(94)90555-x. PMID 7977097
- [Result] Fihn SD, McDonell MB, Diehr P, Anderson SM, Bradley KA, Au DH, Spertus JA, Burman M, Reiber GE, Kiefe CI, Cody M, Sanders KM, Whooley MA, Rosenfeld K, Baczek LA, Sauvigne A. Effects of sustained audit/feedback on self-reported health status of primary care patients. Am J Med. 2004 Feb 15;116(4):241-8. doi: 10.1016/j.amjmed.2003.10.026. PMID 14969652
- [Result] Felker B, Katon W, Hedrick SC, Rasmussen J, McKnight K, McDonnell MB, Fihn SD. The association between depressive symptoms and health status in patients with chronic pulmonary disease. Gen Hosp Psychiatry. 2001 Mar-Apr;23(2):56-61. doi: 10.1016/s0163-8343(01)00127-x. PMID 11313071
- [Result] Smith NL, Chen L, Au DH, McDonell M, Fihn SD. Cardiovascular risk factor control among veterans with diabetes: the ambulatory care quality improvement project. Diabetes Care. 2004 May;27 Suppl 2:B33-8. doi: 10.2337/diacare.27.suppl_2.b33. PMID 15113780
- [Result] Reiber GE, Au D, McDonell M, Fihn SD. Diabetes quality improvement in Department of Veterans Affairs Ambulatory Care Clinics: a group-randomized clinical trial. Diabetes Care. 2004 May;27 Suppl 2:B61-8. doi: 10.2337/diacare.27.suppl_2.b61. PMID 15113785
- [Result] Reiber GE, McDonell MB, Schleyer AM, Fihn SD, Reda DJ. A comprehensive system for quality improvement in ambulatory care: assessing the quality of diabetes care. Patient Educ Couns. 1995 Sep;26(1-3):337-41. doi: 10.1016/0738-3991(95)00741-h. PMID 7494747
- [Result] Au DH, Kivlahan DR, Bryson CL, Blough D, Bradley KA. Alcohol screening scores and risk of hospitalizations for GI conditions in men. Alcohol Clin Exp Res. 2007 Mar;31(3):443-51. doi: 10.1111/j.1530-0277.2006.00325.x. PMID 17295729
- [Result] Fan VS, Reiber GE, Diehr P, Burman M, McDonell MB, Fihn SD. Functional status and patient satisfaction: a comparison of ischemic heart disease, obstructive lung disease, and diabetes mellitus. J Gen Intern Med. 2005 May;20(5):452-9. doi: 10.1111/j.1525-1497.2005.40057.x. PMID 15963172
- [Result] Ohldin A, Young B, Derleth A, McDonell M, Diehr P, Kiefe C, Fihn S. Ethnic differences in satisfaction and quality of life in veterans with ischemic heart disease. J Natl Med Assoc. 2004 Jun;96(6):799-808. PMID 15233490
- [Result] Henderson WG, Demakis J, Fihn SD, Weinberger M, Oddone E, Deykin D. Cooperative studies in health services research in the Department of Veterans Affairs. Control Clin Trials. 1998 Apr;19(2):134-48. doi: 10.1016/s0197-2456(97)00148-7. PMID 9551278
- [Result] Spertus JA, Winder JA, Dewhurst TA, Deyo RA, Prodzinski J, McDonell M, Fihn SD. Development and evaluation of the Seattle Angina Questionnaire: a new functional status measure for coronary artery disease. J Am Coll Cardiol. 1995 Feb;25(2):333-41. doi: 10.1016/0735-1097(94)00397-9. PMID 7829785
- [Result] Bradley KA, McDonell MB, Bush K, Kivlahan DR, Diehr P, Fihn SD. The AUDIT alcohol consumption questions: reliability, validity, and responsiveness to change in older male primary care patients. Alcohol Clin Exp Res. 1998 Nov;22(8):1842-9. doi: 10.1111/j.1530-0277.1998.tb03991.x. PMID 9835306
- [Result] Arterburn DE, McDonell MB, Hedrick SC, Diehr P, Fihn SD. Association of body weight with condition-specific quality of life in male veterans. Am J Med. 2004 Nov 15;117(10):738-46. doi: 10.1016/j.amjmed.2004.06.031. PMID 15541323
- [Result] Fan VS, Bryson CL, Curtis JR, Fihn SD, Bridevaux PO, McDonell MB, Au DH. Inhaled corticosteroids in chronic obstructive pulmonary disease and risk of death and hospitalization: time-dependent analysis. Am J Respir Crit Care Med. 2003 Dec 15;168(12):1488-94. doi: 10.1164/rccm.200301-019OC. Epub 2003 Oct 2. PMID 14525798
- [Result] Fan VS, Au DH, McDonell MB, Fihn SD. Intraindividual change in SF-36 in ambulatory clinic primary care patients predicted mortality and hospitalizations. J Clin Epidemiol. 2004 Mar;57(3):277-83. doi: 10.1016/j.jclinepi.2003.08.004. PMID 15066688
- [Result] Bradley KA, Maynard C, Kivlahan DR, McDonell MB, Fihn SD; Ambulatory Care Quality Improvement Project Investigators. The relationship between alcohol screening questionnaires and mortality among male veteran outpatients. J Stud Alcohol. 2001 Nov;62(6):826-33. doi: 10.15288/jsa.2001.62.826. PMID 11838920
- [Result] Spertus JA, Dewhurst TA, Dougherty CM, Nichol P, McDonell M, Bliven B, Fihn SD. Benefits of an "angina clinic" for patients with coronary artery disease: a demonstration of health status measures as markers of health care quality. Am Heart J. 2002 Jan;143(1):145-50. doi: 10.1067/mhj.2002.119894. PMID 11773925
- [Result] Keeffe B, Subramanian U, Tierney WM, Udris E, Willems J, McDonell M, Fihn SD. Provider response to computer-based care suggestions for chronic heart failure. Med Care. 2005 May;43(5):461-5. doi: 10.1097/01.mlr.0000160378.53326.f3. PMID 15838410